CLINICAL TRIAL: NCT00556023
Title: A Phase 1 Dose Escalation Trial Of CP-675,206 In Combination With Gemcitabine In Patients With Chemotherapy Naive Metastatic Pancreatic Cancer
Brief Title: A Phase 1 Study Testing CP-675,206 In Combination With Gemcitabine In Patients With Previously Untreated, Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3671016
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Pancreatic Cancer
Keywords: interventional; dose-finding
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — tremelimumab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CP-675,206 and gemcitabine (Experimental)
  Interventions: Drug: CP-675,206 and gemcitabine

INTERVENTIONS:
Drug: CP-675,206 and gemcitabine — Escalating doses of CP-675,206 will be administered by IV infusion on day 1 of each 84-day treatment cycles (doses of 6, 10 and 15 mg/kg are planned). Gemcitabine will be administered by IV infusion, at a fixed dose of 1000 mg/m2 on days 1 (prior to CP-675,206) and again on days 8, 15, 29, 36, 43, 57, 64, and 71. Repeated cycles of gemcitabine and CP-675,206 will be administered until patients develop progressive disease or unacceptable toxicity, or for a maximum of 4 cycles, whichever occurs first.

SUMMARY:
The purpose of this study is to determine the safety and tolerability of different doses of CP-675,206 in combination with gemcitabine and to determine the maximum dose of CP-675,206 that is well tolerated when given in combination with gemcitabine to patients with advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic pancreatic cancer
* Patient must have adequate bone marrow, liver and kidney function
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1
* Chemotherapy naive
* Inoperable pancreatic cancer

Exclusion Criteria:

* Patient must not have received prior systemic therapy for pancreatic cancer
* Patient must not have previously received anti-CTLA4 therapy
* History of chronic inflammatory or autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities: assessed through adverse event data collected weekly | 8 week intervals

SECONDARY OUTCOMES:
HAHA Response to CP-675,206: | 12 months
Lymphocyte Subset Analysis: | 12 months
Cytokine Analysis: | 12 months
Pharmacogenomic Analysis: | 1 month
Overall Survival: | 12 months
Pharmacokinetics of CP-675,206 and Gemcitabine: | 2 months
Best Overall Response: | 3 months
Duration of Tumor Response: | 3 months
Progression-Free Survival: | 5 months

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (3):
  - Research Site, Edmonton, Alberta
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Italy (2):
  - Research Site, Candiolo (TO)
  - Research Site, Roma

REFERENCES:
- [Derived] Aglietta M, Barone C, Sawyer MB, Moore MJ, Miller WH Jr, Bagala C, Colombi F, Cagnazzo C, Gioeni L, Wang E, Huang B, Fly KD, Leone F. A phase I dose escalation trial of tremelimumab (CP-675,206) in combination with gemcitabine in chemotherapy-naive patients with metastatic pancreatic cancer. Ann Oncol. 2014 Sep;25(9):1750-1755. doi: 10.1093/annonc/mdu205. Epub 2014 Jun 6. PMID 24907635